CLINICAL TRIAL: NCT02378116
Title: Can We Protect the Brain Against Thrombus Embolism by Closing the Left Atrial Appendage During Open Heart Surgery
Brief Title: Left Atrial Appendage Closure During Open Heart Surgery
Acronym: LAACS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Frederiksberg University Hospital (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Hvidovre University Hospital (Other)
Responsible Party: Principal Investigator, Jesper Park Hansen, MD., Jesper Park Hansen, MD, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: H-3-2010-017
Record Dates: First submitted 2014-09-16; First posted 2015-03-04 (Estimated); Last update posted 2018-02-27 (Actual); Status verified 2018-02

CONDITIONS: Atrial Fibrillation; Cerebral Embolism; Stroke
MeSH Terms: conditions — Atrial Fibrillation; Intracranial Embolism; Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): On the control group is done MRI scans of the brain, and patients can be elected for monitoring and/or bicycle stress test to test for neurohormones.
- Surgical Closure (Active Comparator): During open heart surgery, the surgeon closes the left atrial appendage. The research group recommend a double closure with both a ligation and suture, but a single suture is also accepted.
  Interventions: Procedure: Surgical closure of the left atrial appendage

INTERVENTIONS:
Procedure: Surgical closure of the left atrial appendage — When patients are randomized to surgical closure, the surgeon is informed to close the left appendage. Closure is documented by a member of the research group at the site.
  Arms: Surgical Closure

SUMMARY:
Because atrial fibrillation occurs frequently in heart surgery patients, our overall hypothesis is that systematic closing the left atrial appendage during surgery will reduce cerebral embolism coming from the thrombus formation in the left atrium.

The specific hypothesis which sought tested is that closure of the left atrial appendage in connection with elective CABG and / or valve surgery will lead to fewer strokes and micro cerebral infarcts measured by MRI.

DETAILED DESCRIPTION:
Patients are included prior to surgery. An MRI is performed at baseline. At the day of surgery, patients is randomized to closure/left open left atrial appendage.

During surgery, a maximum of 15 ml blood and a right atrium biopsy are taken for further analyses. Additionally, a biopsy of the left atrium appendage is collected from the group of patients randomized for closure.

The study group recommend a double closure. After discharge a second MRI is performed and the final MRI is performed after a minimum of six months.

The final contact with the patient is done one year after surgery at the earliest. Where a clinical interview is done over the phone and the patients clinical records are screened for cerebral ischaemic events and atrial fibrillation.

During the study period, some patients are elected for a bicycle stress test to test for levels of neurohormones, and some are elected for monitoring with Holter.

There will also be performed transesophageal echocardiography on interested patients in order to test for the quality of surgical closure.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years old.
* elective open heart surgery By-pass (CABG) and/or valve surgery
* signed informed consent

Exclusion Criteria:

* off pump heart surgery
* endocarditis
* Patients with metal implants not suitable for MRI
* Patients with planned implantation of pacemaker after surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2011-10; Primary Completion 2017-01-01 (Actual); Study Completion 2017-01-01 (Actual)

PRIMARY OUTCOMES:
Combined endpoint: Stroke and/or changes in number of micro cerebral infarcts identified with MRI at follow up compared to discharge from surgery. | Endpoint is earliest one year after randomization. Follow-up is continued for the entire length of the study. The rationale for this is that this one intervention provides lifetime protection against ischaemic damage.

OTHER OUTCOMES:
Comparison of increase of Atrial Natriuretic Peptide (ANP) during exercise testing in open versus closed left atrial appendage. 20 Patients have been included and have finished the sub study as of Jan 2015 | Exercise test is scheduled three months after surgery. Blood samples are analyzed and levels of ANP are assessed.
  The investigators want to test if the levels of NT-proANP (pro-hormone of atrial natriuretic peptide) will change during stress in patients with a closed left atrial appendage, compared to the control group. The test is performed on a ergometer-bicycle, with blood samples taken at baseline and after maximum exercise. The levels of neurohormones will then be analyzed.
  The study is done in order to better map of the areas producing neurohormones in the heart.
Study of recurrent atrial fibrillation in patients with per-operative onset. | Between three months and two years after surgery, the patients will be included for a 6-7 days monitoring of heart rhythm. Data last patient will have completed monitoring December 2015
  Patients who develop atrial fibrillation after surgery, with no previous history of atrial fibrillation, and who are discharged in sinus rhythm, will be offered monitoring of heart rhythm with Holter monitor. Preferably for one week, in order to investigate, weather restoring sinus rhythm is permanent, or if debut of atrial fibrillation is onset of a new disease more than a symptom form surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Jesper P. Hansen, MD, Study Director — University of Copenhagen
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

REFERENCES:
- [Derived] Madsen CV, Park-Hansen J, Holme SJV, Irmukhamedov A, Carranza CL, Greve AM, Al-Farra G, Riis RGC, Nilsson B, Clausen JSR, Norskov AS, Kruuse C, Truelsen TC, Dominguez H. Randomized Trial of Surgical Left Atrial Appendage Closure: Protection Against Cerebrovascular Events. Semin Thorac Cardiovasc Surg. 2023 Winter;35(4):664-672. doi: 10.1053/j.semtcvs.2022.06.012. Epub 2022 Jun 28. PMID 35777693
- [Derived] Park-Hansen J, Holme SJV, Irmukhamedov A, Carranza CL, Greve AM, Al-Farra G, Riis RGC, Nilsson B, Clausen JSR, Norskov AS, Kruuse CR, Rostrup E, Dominguez H. Adding left atrial appendage closure to open heart surgery provides protection from ischemic brain injury six years after surgery independently of atrial fibrillation history: the LAACS randomized study. J Cardiothorac Surg. 2018 May 23;13(1):53. doi: 10.1186/s13019-018-0740-7. PMID 29792215